CLINICAL TRIAL: NCT01396863
Title: Acute Brain Volume Changes in Haemodialysis: Comparison of Low Flux Haemodialysis With Pre-dilution Haemodiafiltration
Brief Title: Brain Swelling During Dialysis
Acronym: BRASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VEK20100228
Record Dates: First submitted 2011-07-13; First posted 2011-07-19 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: End Stage Renal Disease
Keywords: Renal dialysis; Hemodiafiltration; Hemodialysis; MRI
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First treatment HDF (Active Comparator): The patient will receive treatment with pre-dilution hemodiafiltration during the first examination day. During the second examination day the patient will receive treatment with low flux hemodialysis.
  Interventions: Procedure: HDF during the first examination
- First treatment HD (Active Comparator): The patient will receive treatment with low flux hemodialysis during the first examination day. During the second examination day the patient will receive treatment with pre-dilution hemodiafiltration.
  Interventions: Procedure: HD during the first examination

INTERVENTIONS:
Procedure: HDF during the first examination — The patient will receive treatment with pre-dilution hemodiafiltration during the first examination.
  During the second examination the patient will receive treatment with low flux hemodialysis.
  MRI of the brain will be performed before and after the treatment. The MRI-data will later be processed to determine the degree of brain volume change due to the treatment.
  Arms: First treatment HDF
Procedure: HD during the first examination — The patient will receive treatment with low flux hemodialysis during the first examination.
  During the second examination the patient will receive treatment with pre-dilution hemodiafiltration.
  MRI of the brain will be performed before and after the treatment. The MRI-data will later be processed to determine the degree of brain volume change due to the treatment.
  Arms: First treatment HD

SUMMARY:
The proposed controlled, randomized study aims to compare pre-dilution hemodiafiltration (HDF) and low flux hemodialysis (HD) regarding acute changes in the brain.

The study consist of two examination days placed one week apart. 12 HD patients will be recruited to the study. The patients will be randomly placed in two groups: Pre-dilution hemodiafiltration during the first examination and low flux hemodialysis during the second day or vice versa.

Brain Magnetic Resonance Imaging (MRI) will be obtained before and after both treatments. The MRI-data will later be processed to estimate brain volume changes during the two types of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed consent
* Patient with end-stage renal disease (ESRD)
* Stabile hemodialysis treatment (Kt/V ≥ 1.3)
* No contraindications against MRI (pacemaker or other metal implants, claustrophobia, severe adiposity)
* Weight <140kg

Exclusion Criteria:

* Clinical signs of new structural, thromboembolic or vascular brain disease the last 3 month before entering the study
* Changes in corticosteroid treatment during the last two weeks
* Change in diuretics during the last two weeks
* Non-compliant with regard to salt and fluid intake
* Acute disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Percent Brain Volume Change (PBVC) | Brain volume before and after one hemodialysis session (4,5 hours) and one session of hemodiafiltration (4,5 hours). Dialysis sessions are performed one week apart.
  Brain volume before and after one hemodialysis session (4,5 hours) and one session of hemodiafiltration (4,5 hours). Dialysis sessions are performed one week apart. Randomization determines the order of treatment (hemodialysis vs hemodiafiltration).
  MRI-data will later be processed to estimate the PBVC.

CONTACTS AND LOCATIONS:
Overall Officials: Jens D. Jensen, MD, PhD, Study Director — Department of Renal Medicine C, Aarhus University Hospital, Skejby, Denmark; Niels Johansen, BSc Medicine, Principal Investigator — Department of Renal Medicine C, Aarhus University Hospital, Skejby, Denmark
Locations (2):
- Denmark (2):
  - Department of Renal Medicine C, Aarhus University Hospital, Skejby, Aarhus N
  - The MR-Research Centre, Aarhus University Hospital, Skejby, Aarhus N

REFERENCES:
- [Derived] Kulkarni M, Prabhu AR, Rao IR, Nagaraju SP. Interventions for preventing haemodialysis dysequilibrium syndrome. Cochrane Database Syst Rev. 2024 May 22;5(5):CD015526. doi: 10.1002/14651858.CD015526.pub2. PMID 38775299